CLINICAL TRIAL: NCT05033912
Title: An Open-Label Ascending Single-Dose, and Randomized, Double-blind, Placebo-controlled, Ascending Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CST-2032 in Healthy Volunteers and Subjects With Mild Cognitive Impairment or Parkinson's Disease
Brief Title: A Study of CST-2032 in Subjects With Cognitive Impairment
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: CuraSen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CST2032-CLIN-007
Record Dates: First submitted 2021-08-24; First posted 2021-09-05 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Mild Cognitive Impairment (MCI); Parkinson Disease (PD)
MeSH Terms: conditions — Cognitive Dysfunction; Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This is a phase1, randomized sequence of placebo, low-, mid- and high-dose CST-2032 after a pre-administered dose of 3 mg CST-107.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Sequence 1 (Experimental): Subjects will receive daily doses of matching placebo for CST-2032 and CST-107 on Day 1, 1mg CST-2032 & 3mg CST-107 on Day 2, 3mg CST-2032 & 3mg CST-107 on Day 3, & 9mg CST-2032 and 3mg CST-107 on Day 4.
  Interventions: Drug: CST-2032, matching placebo for CST-2032, CST-107
- Treatment Sequence 2 (Experimental): Subjects will receive daily doses of 1mg CST-2032 & 3mg CST-107 on Day 1, 3mg CST-2032 & 3mg CST-107 on Day 2, & 9mg CST-2032 and 3mg CST-107 on Day 3, and matching placebo for CST-2032 and CST-107 on Day 4.
  Interventions: Drug: CST-2032, matching placebo for CST-2032, CST-107
- Treatment Sequence 3 (Experimental): Subjects will receive daily doses of 3mg CST-2032 & 3mg CST-107 on Day 1, & 9mg CST-2032 and 3mg CST-107 on Day 2, matching placebo for CST-2032 and CST-107 on Day 3, and 1mg CST-2032 & 3mg CST-107 on Day 4.
  Interventions: Drug: CST-2032, matching placebo for CST-2032, CST-107
- Treatment Sequence 4 (Experimental): Subjects will receive daily doses of 9mg CST-2032 and 3mg CST-107 on Day 1, matching placebo for CST-2032 and CST-107 on Day 2, 1mg CST-2032 & 3mg CST-107 on Day 3, and 3mg CST-2032 & 3mg CST-107 on Day 4.
  Interventions: Drug: CST-2032, matching placebo for CST-2032, CST-107

INTERVENTIONS:
Drug: CST-2032, matching placebo for CST-2032, CST-107 — CST-2032 and matching placebo oral liquid; CST-107 white capsules

SUMMARY:
This study will evaluate the effects of CST-2032 when administered with pre-administered CST-107 on safety, tolerability, cognition, cerebral perfusion, and cerebral metabolism in patients with cognitive impairment.

DETAILED DESCRIPTION:
This is a phase1, randomized sequence of placebo, low-, mid- and high-dose CST-2032 in Subjects with cognitive impairment. Sixteen (16) subjects with cognitive impairment will be enrolled. The first subject enrolled will be dosed as a sentinel. If no significant safety issues are noted in the sentinel subject, the remaining subjects will be dosed starting 24 hours after the Day 4 dose for the sentinel subject.

Subjects will have the option to attend all study visits as outpatients or be admitted for a 4-5-night confinement period at the research facility. Subjects will receive matching placebo for CTS-2032, 1mg, 3mg, and 9 mg CST-2032 two hours after a pre-administered dose of 3 mg CST-107 in a randomized sequence on Days 1, 2, 3 and 4.

Cognitive assessments (CANTAB) and a verbal fluency test will be administered daily. If operationally feasible, subjects will also undergo arterial spin labeling (ASL) magnetic resonance (MRI) imaging of the brain on Days 1 and 4.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 45-75 years at the time of informed consent.
* Unless confirmed to be azoospermic (vasectomized or secondary to medical cause), males must agree to use a male condom plus partner use of an additional contraceptive method from the start of confinement or Day -1 up to 90 days after the last study drug administration when having penile-vaginal intercourse with a woman of childbearing potential who is not currently pregnant. Sperm donation is not allowed during this period. Note: Men with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a condom during each episode of penile-vaginal penetration.
* Females of childbearing potential must have a negative serum pregnancy test during Screening and a negative urine pregnancy test before first dose of study drug. In addition, they must be willing to abstain from egg collection or donation from start of Screening through 90 days after the last study drug administration.
* Females of childbearing potential (i.e., not postmenopausal or surgically sterile) who have a male partner must agree to one of the following options from signing of informed consent through 90 days after the last study drug administration: use of a highly effective method of birth control, or confirmed sterilization of a monogamous partner, or practice abstinence.
* Females of non-childbearing potential may be enrolled if they are postmenopausal or have documented evidence of surgical sterilization.
* Stable medical conditions for at least 3 months prior to Screening visit (e.g., hypertension, dyslipidemia)
* Stable use of vitamin E (up to 400 IU daily), estrogens, aspirin (75-300 mg daily), blood pressure medications (except for adrenergic agents), and cholesterol-lowering agents for at least 3 months prior to screening is allowed.
* In generally good health based on medical and surgical history, BMI, physical examination, vital signs, 12-lead ECG and laboratory values, including hematology and chemistry values.
* Clinical laboratory values within normal limits or, if abnormal, must be judged to be clinically insignificant.
* Able to understand and sign the written Informed Consent Form (ICF).
* Willing to follow the protocol requirements and comply with protocol restrictions.

In addition, for subjects with MCI:

* Must meet the criteria for amnestic Mild Cognitive Impairment (MCI), as per the National Institute on Aging-Alzheimer's Association core clinical criteria.
* No dementia according to International Classifications of Diseases (ICD)-10 and Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV.
* A score of greater than or equal to one standard deviation below age and educational norms in the Digit Symbol Substitution Test (DSST) during screening.
* A memory complaint reported by the subject or his/her partner.
* Cognitive decline not primarily caused by vascular, traumatic, or medical problems.
* Preserved basic activities of daily living and no more than minimal impairment.

In addition, for subjects with PD:

* Parkinson's disease (PD) defined by the cardinal sign, bradykinesia, plus the presence of at least 1 of the following: resting tremor, rigidity, or impairment of postural reflexes, and without any other known or suspected cause of Parkinsonism
* Modified Hoehn & Yahr stage ≤ 3 during "On" period as documented in the 3 months prior to Screening.
* Mini Mental Status Examination (MMSE) score ≥26.
* If taking medications for PD, subjects on stable (≥3 months prior to Day 1) levodopa/carbidopa or levodopa/benserazide, monoamine oxidase type B inhibitors, dopamine agonists or catechol-O-methyltransferase inhibitors are allowed. Subjects on β-antagonists are not allowed.

Exclusion Criteria:

* Female subjects who are pregnant or lactating.
* History of any significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, metabolic, psychological, or musculoskeletal disease.
* Subjects with a history of malignant disease, including solid tumours and hematologic malignancies (except basal cell and squamous cell carcinomas of the skin that have been completely excised and are considered cured).
* Calculated creatinine clearance of ≤60 mL/min.
* Positive screening test for human immunodeficiency virus (HIV).
* Positive screening test for hepatitis C antibody (HCV Ab) or current hepatitis B infection (defined as positive for hepatitis B surface antigen [HBsAg] at Screening). Subjects with immunity to hepatitis B (defined as negative HBsAg and positive hepatitis B core antibody [anti-HBc]) are eligible to participate in the study.
* Positive test for and current infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at Screening, or evidence of possible ongoing infection based on body temperature (> 37.3 oC), blood oxygen (<90 %) at the start of first confinement or Day -1.
* History of epilepsy, seizure disorder or any unexplained black-outs.
* Suicidal ideation with actual intent or plan ("Yes" answer on the Columbia-Suicide Severity Rating Scale [C-SSRS] ideation items 4 or 5) within 3 months prior to study Screening.
* History of drug or alcohol abuse ≤12 months prior to Screening.
* History of tobacco use including cigarettes, cigars, vapes or e-cigarettes ≤6 months prior to Screening.
* A positive test for drugs of abuse, cotinine or alcohol during Screening or prior to dosing.
* Unwilling or unable to abstain from alcohol or caffeine for 48 hours prior to dosing until end of each confinement or dosing period.
* Current use of any prohibited medication, over-the-counter medication, or herbal supplements/products.
* History of relevant cardiovascular disease including angina, hypertension (unless currently under control with stable medications), heart failure, coronary insufficiency, cardiac arrhythmias, diabetes mellitus, hyperthyroidism, convulsion disorders, bronchial asthma, clinically significant sinus bradycardia and greater than first degree conduction block.
* Clinically significant abnormal clinical laboratory test values.
* Clinically significant abnormalities in 12-lead ECG, including marked baseline prolongation of QT/QTcF interval (e.g., repeated demonstration of a QTcF interval >450 msec) at Screening.
* Prior treatment with any investigational drug ≤30 days prior to dosing (Day 1), or ≤5 half-lives of the drug (whichever is longer), or current enrolment in any other study treatment or disease study.
* Vaccinations ≤14 days prior to dosing.
* Donation or loss of ≥500 mL of blood or plasma within 30 days prior to dosing.
* Inability to undergo a clinical MRI of the brain without contrast.
* Clinically significant brain abnormalities based on T1 weighted MRI during screening.
* Any other reason which prompts the Principal Investigator to consider that it is not in the best interest of the subject to participate in the study.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events | Day -1, Days 1-4 of the treatment period
  The number of subjects experiencing treatment-emergent adverse events after receiving CST-2032 doses of 1mg, 3mg and 9mg compared to placebo
Vital Signs | Day -1, Days 1-4 of the treatment period
  Change from Baseline in supine blood pressure (diastolic blood pressure and systolic blood pressure) after CST-2032 doses of 1mg, 3mg, and 9mg compared to placebo
Electrocardiograms (ECGs) | Day -1, Days 1-4 of the treatment period
  Change from Baseline in QTc interval using the Fredericia (QTcF) and Bazett (QTcB) corrections after CST-2032 doses of 1mg, 3mg, and 9mg compared to placebo

SECONDARY OUTCOMES:
Change from Baseline in CANTAB Reaction Time Task | Day -1, Days 1-4 of the treatment period
  Measures changes in cognition by testing psychomotor speed (selecting a flashing circle on a touch tablet screen as quickly as possible).
Change from Baseline in CANTAB Paired Associates Learning Test | Day -1, Days 1-4 of the treatment period
  Measures changes in cognition by testing attention (remembering the location of an abstract pattern on a touch tablet screen).
Change from Baseline in CANTAB Verbal Recognition Memory | Day -1, Days 1-4 of the treatment period
  Measures changes in cognition by testing memory (recall of 18 words flashed onto a touch tablet screen).
Change from Baseline in CANTAB Rapid Visual Information Processing | Day -1, Days 1-4 of the treatment period
  Measures changes in cognition by testing sustained attention, response accuracy, target sensitivity and reaction times. Single digits appear in random order in the center of a touch tablet screen and subjects must detect a series of 3-digit target sequences and respond by touching the button at the bottom of the screen when they see the final number of the sequence.
Change from Baseline in CANTAB Adaptive Tracking Task | Day -1, Days 1-4 of the treatment period
  Measures changes in visual and motor coordination and vigilance. In this task, a small circle (target) continuously moves across the screen in a semi-randomized fashion, so as to minimize the subject's ability to predict the trajectory of the target. The subject is instructed to use his/her finger on the touch screen to move a small dot so that it is consistently within the center of the moving target on the screen. During the test, the speed of the circle is adjusted in response to the subject's ability to keep the dot in the circle, ensuring that the test is adapted to the individual subject.
Change from Baseline in Verbal Fluency Test | Day -1, Days 1-4 of the treatment period
  Measures changes in cognition by assessing executive function, and requires the generation of words from initial letters or belonging to a specific category under a time constraint. Subjects are given 1 minute to say aloud as many words they can think of that begin with the letter F, avoiding repetitions or the same words with different endings. The total score is the number of correct words generated. Subjects are also given 1 minute to say aloud as many animals they can think of, avoiding repetitions. The total score is the number of animals generated.
Change from Baseline in ASL MRI scans of the brain | Pre- and Post-dose on Days 1 and 4
  Measures cerebral blood flow (CBF). CBF is defined as the volume of blood delivered to a given mass of brain tissue in a given time.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — CuraSen Therapeutics, Inc.

IPD SHARING:
Plan to Share IPD: No